CLINICAL TRIAL: NCT01564433
Title: The Effects of an Electromechanical Gait Trainer in Gait Impairments and Endurance in Patients With Cerebral Palsy: a Randomized Control Trial
Brief Title: Effects of Electromechanical Gait Trainer in Patients With Cerebral Palsy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Prof. Smania Nicola, Universita di Verona
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PCI-GT-2
Record Dates: First submitted 2012-03-14; First posted 2012-03-27 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Cerebral Palsy
Keywords: robotics; rehabilitation; gait; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gait trainer treatment (Experimental)
  Interventions: Procedure: Device: Electromechanical gait trainer
- Conventional group (Active Comparator)
  Interventions: Procedure: Convetional control treatment

INTERVENTIONS:
Procedure: Device: Electromechanical gait trainer — The experimental group will be subjected to 12-30 minute session (3 per week: Monday, Wednesday, Friday) of repetitive locomotor therapy on the Gait Trainer (Reha-Stim, Berlin, Germany), followed by 20 minutes of passive joint mobilization and stretching exercises. The GT-I consists of a double crank and rocker gear system, composed of two footplates positioned on two bars (coupler), two rockers, and two cranks that provide the propulsion. While using the gait trainer, individuals are secured in a harness and positioned on two footplates, whose movements simulate stance and swing phase, with a ratio of 60% to 40% between the two phases. The body weight was initially reduced by 30% and then progressively increased.
  Arms: Gait trainer treatment
Procedure: Convetional control treatment — The control group will be subjected to a conventional treatment that will consist of three different sets of exercises: 1) passive joint mobilization and stretching of lower limb muscles; 2) muscle strengthening exercises; 3) gait exercises. Each set of exercises lasted 10, 15 and 15 min, respectively with 2,5 min at rest between each set for a total of 40 minutes.
  Arms: Conventional group

SUMMARY:
Cerebral Palsy (CP) describes a group of chronic conditions affecting body movement and muscle coordination caused by damage to one or more areas of the brain, usually occurring during fetal development or infancy. One of the most disabling mobility impairments in CP is gait impairment, clinically characterized by reduced speed and endurance, as well as reduced step, stride length and toe clearance during gait.

Recently, gait rehabilitation methods in patients with neurological impairment have relied on technological devices, which drive the patient's gait in a body-weight support condition and emphasize the beneficial role of repetitive practice. Early studies in gait rehabilitation in patients with CP were carried out by using partial body-weight support treadmill training (PBWSTT) and robotic-assisted treadmill therapy. Despite their potential, these technologies have practical limitations in their routine application.

More recently, several studies have focused on the use of a new electromechanical gait trainer (Gait Trainer GT I; Reha-Stim, Berlin, Germany) in adult patients who have experienced a stroke. They have shown that training with this device may significantly improve gait performance. Despite the clinical impact of this new rehabilitative procedure, to date, no studies have been conducted on its use in children with CP.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) describes a group of chronic conditions affecting body movement and muscle coordination caused by damage to one or more areas of the brain, usually occurring during fetal development or infancy. The motor disorders of CP are often accompanied by disturbances of sensation, cognition, communication, perception, behavior, and/or a seizure disorder. One of the most disabling mobility impairments in CP is gait impairment, clinically characterized by reduced speed and endurance, as well as reduced step, stride length and toe clearance during gait.

Recently, gait rehabilitation methods in patients with neurological impairment have relied on technological devices, which drive the patient's gait in a body-weight support condition and emphasize the beneficial role of repetitive practice. The rationale for these approaches originates from animal studies which have shown that repetition of gait movements may enhance spinal and supraspinal locomotor circuit.

Early studies in gait rehabilitation in patients with CP were carried out by using partial body-weight support treadmill training (PBWSTT) and robotic-assisted treadmill therapy. The majority of these studies consisted of single case, small or unselected patient samples and/or uncontrolled trials. In a recent randomized control trial study, Willoughby et al. showed that PBWSTT was no more effective than overground walking for improving walking speed and endurance in children with CP. They concluded that the progressive reduction of body weight support along with adding concurrent overground walking practice to a treadmill training protocol may increase the intensity of training and assist with carry over of improvements to overground walking. Despite their potential, these technologies have practical limitations in their routine application: PBWSTT requires the assistance of one or two physiotherapists to control the patient's weight shift and lower limb position during training and proper placement of the patient onto the machine (Lokomat, Hokoma Inc., Volketswill, Switzerland) for robotic-assisted treadmill training is time-consuming.

More recently, several studies have focused on the use of a new electromechanical gait trainer (Gait Trainer GT I; Reha-Stim, Berlin, Germany) in adult patients who have experienced a stroke. They have shown that training with this device may significantly improve gait performance. Despite the clinical impact of this new rehabilitative procedure, to date, no studies have been conducted on its use in children with CP.

The primary aim of the present randomized controlled trial is to evaluate whether repetitive locomotor training with the Gait Trainer GT I can improve endurance in tetra- or diplegic ambulatory children with CP. The secondary aim was to assess whether training can also have a positive impact on spatiotemporal gait parameters and quality of life.

Study Design Randomised controlled, blinded clinical trial.

Materials and methods Twenty CP patients will be enrolled in the study. The inclusion criteria will be: bilateral lower limb (diplegic or tetraplegic) CP, 10 to 18 years of age, GMFCS levels II to IV, walk by themselves or with the use of an assistance device for at least 10 meters, maintain a sitting position without assistance and follow instructions and participate in the rehabilitative program. The exclusion criteria will be: lower limb spasticity >2 on the Modified Ashworth Scale, severe lower limb contractures, cardiovascular diseases, orthopedic surgery or neurosurgery in the past 12 months or Botulinum toxin and injections within 6 months before the beginning of the study.

At the moment of recruitment (before treatment), at the end of treatment (6 weeks) and one month and two months after the end of the treatment (FU) each patient will be tested with the following clinical and instrumental procedures. Clinical assessment procedures: 6-minute Walking Test, Ten Meter Walking Test, Gross Motor Classification System, Child Health Questionnaire (CHQ-PF50) Italian version, Wee FIM and Energy Expenditure Index. Instrumental assessment procedures: Gait analysis by means of GAITRite® System and measure of energy cost by COSMED K4b2.

As primary outcome measure will be considered the 6-minute Walking Distance Test. As secondary outcomes measures will be considered Ten Meter Walking Test, Gross Motor Classification System, Child Health Questionnaire (CHQ-PF50) Italian version, Wee FIM and Energy Expenditure Index, Spatio-temporal parameter with GAITRite® System and measure of energy cost by COSMED K4b2. The allocation in the two groups will be done with simple randomisation.

Patients will be randomized into two groups. The first group (experimental group) will be subjected to 12 treatment session (3 sessions/week) on Gait Trainer machine for one month. The second group (control group) will undergo to a conventional treatment with the same duration and frequency of the experimental group. Data will be analysed by means parametric and non-parametric tests. Both, within and between groups comparison will be performed. Data will be analyzed using SPSS software (ver 11.0; SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* bilateral lower limb (diplegic or tetraplegic) Cerebral Palsy
* 10 to 16 years of age
* GMFCS levels II to IV
* walk by themselves or with the use of an assistance device for at least 10 meters
* maintain a sitting position without assistance
* follow instructions and participate in the rehabilitative program

Exclusion Criteria:

* lower limb spasticity >2 on the Modified Ashworth Scale
* severe lower limb contractures
* cardiovascular diseases
* orthopedic surgery or neurosurgery in the past 12 months or Botulinum toxin injections within 6 months before the beginning of the study

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Six Minute Walking Test | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  The patient will be asked to walk at her/his self-selected walking speed in the gym along during the instrumental test.

SECONDARY OUTCOMES:
Ten Meter Walking Test | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
  This is a validated test for the clinical evalua- tion of walking speed.21 The subject will be asked to walk at her/his self-selected walking speed along the central 10 m of a 14-m linoleum-covered walkway. A digital stopwatch will be used to time the walks.
Wee FIM | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
  This widely used scale for the evaluation of disability in children with CP investigates three main domains: self-care, mobility, and cognition (score, 18Y126; high, best performance).
Spatio-temporal gait analysis | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
  Spatio-temporal gait analysis will be evaluated by using a computerized system called GAITRite system (Gold, version 3.2 b - CIR Systems, Inc, Havertown, PA). Patients will ask to ambulate along the 7.66m electronic walkway at their fastest speed. The following gait parameters will be considered: gait speed (cm/sec), cadence (step/min), stride length (cm), step length (cm), heel to heel base support (cm), swing of cycle (%), stance of cycle (%), single support of cycle (%) and double support of cycle (%)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fiaschi, Professor, Study Chair — Department Neurological, Neuropsychological, Morphological and Movement Sciences, University of Verona, Verona, Italy
Locations (1):
- S.S.O. di Riabilitazione dell'Ospedale Policlinico, Verona, Italy

REFERENCES:
- [Background] Willoughby KL, Dodd KJ, Shields N, Foley S. Efficacy of partial body weight-supported treadmill training compared with overground walking practice for children with cerebral palsy: a randomized controlled trial. Arch Phys Med Rehabil. 2010 Mar;91(3):333-9. doi: 10.1016/j.apmr.2009.10.029. PMID 20298820
- [Background] Borggraefe I, Schaefer JS, Klaiber M, Dabrowski E, Ammann-Reiffer C, Knecht B, Berweck S, Heinen F, Meyer-Heim A. Robotic-assisted treadmill therapy improves walking and standing performance in children and adolescents with cerebral palsy. Eur J Paediatr Neurol. 2010 Nov;14(6):496-502. doi: 10.1016/j.ejpn.2010.01.002. Epub 2010 Feb 6. PMID 20138788
- [Background] Willoughby KL, Dodd KJ, Shields N. A systematic review of the effectiveness of treadmill training for children with cerebral palsy. Disabil Rehabil. 2009;31(24):1971-9. doi: 10.3109/09638280902874204. PMID 19874075
- [Background] Damiano DL, DeJong SL. A systematic review of the effectiveness of treadmill training and body weight support in pediatric rehabilitation. J Neurol Phys Ther. 2009 Mar;33(1):27-44. doi: 10.1097/NPT.0b013e31819800e2. PMID 19265768
- [Background] Foley A, Horwood J, Hall R. Language for change. Aust Fam Physician. 1980 Jun;9(6):416-22. No abstract available. PMID 7213237